CLINICAL TRIAL: NCT06667934
Title: Clinical Trial of Zuoqing SAN in Treating Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Heng Deng, Dr., The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024AH-98-01; 2021AH9987 (Other: Anhui Province key specialist project)
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Zuoqing powder was dissolved in 100ml normal saline, retained enema, once a night
  Interventions: Drug: Zuoqing powder was dissolved in 100ml normal saline, retained enema, once a night
- Control Group (Active Comparator): Methalazine supposers anal once a day
  Interventions: Drug: Methalazine suppository was given rectally once a day

INTERVENTIONS:
Drug: Zuoqing powder was dissolved in 100ml normal saline, retained enema, once a night — Zuoqing powder was dissolved in 100ml normal saline, retained enema, once a night
  Other Names: retained enema with Zuoqing powder , once a night
  Arms: Study Group
Drug: Methalazine suppository was given rectally once a day — Methalazine suppository was given rectally once a day
  Arms: Control Group

SUMMARY:
The exact efficacy of Zuoqing SAN enema in the treatment of Ulcerative colitis (UC) has been clinically verified. In this study, Zuoqing SAN was used to treat UC patients with large intestine damp-heat syndrome, and the traditional chinese medicine (TCM) syndrome type was large intestine damp-heat syndrome. The changes of symptoms and signs of patients before and after treatment were observed and compared, and the clinical efficacy of Zuoqing SAN in the treatment of UC large intestine damp-heat syndrome was evaluated by combining the changes of patients' symptoms, related blood indicators, improved Mayo total score, overall syndrome efficacy, clinical comprehensive efficacy and other aspects. By replicating the rat UC model, the effects of Zuoqing SAN on general survival state, colonic gross appearance and histopathological changes, related inflammatory factors, peroxisome proliferator-activated receptor γ (PPAR-γ) /nuclear factor kappa-B（NF-κB) /signal transducerand activator of transcription 1 (STAT1) pathway, macrophage M1, M2 phenotype and microangiogenesis were observed in UC rats. Thus, the specific mechanism of Zuoqing SAN in the treatment of UC was revealed. In this study, the therapeutic effect of Zuoqing Powder on UC was investigated through clinical and animal experiments, and the specific mechanism of action was studied.

ELIGIBILITY:
Inclusion Criteria:① Clinically diagnosed UC; ② The severity of UC is mild to moderate.

-

Exclusion Criteria:① The severity of UC is severe; ②patient with Severe liver, kidney, heart and brain diseases; ③ Patients with Chinese medicine allergy; ④ Pregnant or lactation patients.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms: frequency of stool | Follow-up for 6 months
  Symptoms: frequency of stool in one day, or Daily number of bowel movements

IPD SHARING:
Plan to Share IPD: Yes
We can share IPD with other researchers. When our research results are phased, other research groups can watch and participate in the discussion of the research plan.